CLINICAL TRIAL: NCT02239653
Title: Randomized Controlled Trial to Reduce Calorie Intake From Sugar-sweetened Beverages by Children 1 - 12 Years of Age
Brief Title: Reduction of Excessive Calories From Beverages in Children
Acronym: MWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201403027
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Unhealthy Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physician communication (Experimental): The "Milk. Water. Period" intervention comprises brochures, posters, and key talking points for use by primary pediatricians to use in discussion with the parent about the child's beverages consumption.
  Interventions: Behavioral: Physician communication
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Physician communication
  Arms: Physician communication

SUMMARY:
Objective: to test the hypothesis that an intervention comprised of targeted physician and print messages can influence parents to reduce the amount of sugar-sweetened beverages (SSB) and fruit juice they give to their children 1 - 12 years of age.

DETAILED DESCRIPTION:
The study will be conducted through a practice-based research network of community pediatric practices. Participating sites will be randomized to the intervention or control condition (usual care) using a pre-specified randomization scheme derived using computer generated random numbers. The intervention sites will participate in a 30-minute training for using the "Milk. Water. Period" intervention (brochures, posters, key talking points and phone messages) in their office. The goal is for them to discuss beverage consumption and encourage "Milk. Water. Period" for all children 12 months to 12 years old (not yet reached their 13th birthday) at their checkup visit. The primary care provider (PCP) will use the talking points to facilitate the discussion about drink milk and water only and will give a brochure to each family. Assessments will be by telephone interview of the parent 2 to 4 weeks after a check-up visit for the index child.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child age 12 months to 12 years attending for a check-up visit during the study period

Exclusion Criteria:

* Cannot speak English
* No phone access
* Already completed the survey for another child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2014-11-21 (Actual); Study Completion 2014-11-21 (Actual)

PRIMARY OUTCOMES:
Excessive calories from beverages | 2-4 weeks after check-up visit
  percent of children consuming >200 calories/day from soda, SSBs, and fruit juice beverages

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No